CLINICAL TRIAL: NCT00270673
Title: Early Lactate-Directed Therapy on the ICU: A Randomized Controlled Trial
Brief Title: Early Lactate-Directed Therapy in the Intensive Care Unit (ICU)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Medical Center Rijnmond Zuid, Rotterdam (Unknown); Sint Franciscus Gasthuis (Other); Reinier de Graaf Groep (Other); Albert Schweitzer Hospital, Netherlands (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-334
Record Dates: First submitted 2005-12-23; First posted 2005-12-28 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Tissue Hypoxia; Hyperlactatemia
Keywords: Lactate; Tissue hypoxia; Intensive care; Goal- directed therapy
MeSH Terms: conditions — Hyperlactatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Early lactate-directed therapy

SUMMARY:
Blood lactate levels have long been related to tissue hypoxia, a severe condition in critically ill patients associated with the development of organ system failure and subsequent death. Increased blood lactate levels and failure to normalize blood lactate levels during treatment have been associated with increased morbidity and mortality. However, evidence of improved clinical outcome of lactate-directed therapy is limited and difference in the use of blood lactate monitoring in the intensive care unit exists between hospitals. This warrants a study on the efficacy of early blood lactate-directed therapy. In this study the efficacy of 8 hours of early lactate-directed therapy (therapy aimed at resolving tissue hypoxia that is guided by serial blood lactate levels) will be compared with 8 hours of control group therapy (without lactate measurement).

DETAILED DESCRIPTION:
Tissue hypoxia can be defined as a state in which tissue oxygen demand is not met by tissue oxygen delivery (DO2). The presence and persistence of tissue hypoxia is related to the development of organ system failure and subsequent death. However, definite clinical indicators of tissue hypoxia are lacking. In experimental conditions, a mismatch between oxygen delivery and oxygen demand, resulting from either a progressive decrease of any of the components of oxygen delivery (hemoglobin level, arterial oxygen saturation and cardiac output) or an increase in oxygen demand, leads to increases in blood lactate levels. However, as lactate is a normal end product of metabolism, other processes not related to tissue hypoxia have also been linked to increases in blood lactate levels. In clinical conditions increased blood lactate levels and a failure to normalize blood lactate levels during treatment have been associated with increased morbidity and mortality. Even in hemodynamically stable patients with hyperlactatemia, a condition referred to as compensated shock or occult hypoperfusion, lactate levels are related to morbidity and mortality. In our retrospective pilot study, performed in the general ICU of the Erasmus MC (n= 931), we found 40% mortality in patients with blood lactate levels of 3 mmol/l or higher in the early hours of ICU admission. Blow at al. implemented a treatment protocol to increase oxygen delivery, guided by blood lactate levels, in hemodynamically stable trauma patients with occult hypoperfusion. Failure to correct hyperlactatemia after lactate-directed therapy correlated with increased mortality. Rossi et al. studied lactate-directed therapy in children undergoing congenital heart surgery. However, while showing a reduction in morbidity and mortality, they used a historical control group. Only one randomized controlled trial has been performed evaluating lactate-directed therapy. This study of Polonen et al. showed a decrease in morbidity and length of stay in post-cardiac surgery patients using lactate < 2mmol/l (and mixed venous oxygen saturation [SvO2] > 70%) as goals of therapy. Thus, a relevant body of clinical evidence does not yet support routine monitoring of blood lactate levels and lactate-directed therapy in all critically ill patients. As some investigators have even posed strong arguments that increased blood lactate levels are not related to the presence of tissue hypoxia in critically ill patients, some clinicians use increased blood lactate levels to guide therapy whereas others hardly measure lactate levels. The limited evidence of efficacy and the variable clinical use of blood lactate monitoring in different hospitals thus warrants a study on the clinical efficacy of blood lactate monitoring and blood lactate-directed therapy in the ICU.

In general a monitor cannot influence outcome without an associated treatment protocol to guide treatment. We will therefore study the clinical efficacy of repeated blood lactate measurements in combination with a predefined treatment protocol (aimed at resolving tissue hypoxia) during the first hours of intensive care treatment. This pragmatic approach and also the early timing of the intervention are supported by the study of Rivers et al., in which optimizing the balance between oxygen delivery and demand early in the treatment of patients with severe sepsis and septic shock resulted in a 16% absolute mortality reduction.

The pre-defined treatment protocol will consist of components to

1) reduce oxygen demand, 2) increase oxygen delivery and to 3) recruit the microcirculation.

1. Reduction of metabolic oxygen demand has been successfully accomplished by preventing hyperthermia, adequate analgesia or sedation, and mechanical ventilation.
2. Increasing oxygen delivery can be achieved by increasing any of the components of oxygen transport (arterial oxygen saturation, cardiac output and hemoglobin level). However, the oxygen delivering capabilities of stored red blood cells have been debated and adverse effects of red blood cell transfusion have been reported. Best evidence suggests a restrictive transfusion policy in the ICU (transfusion threshold 4.34 mmol/l) with an exception of severe ischemic cardiac disease.
3. Administration (after intravascular volume resuscitation) of nitroglycerin, reverses microcirculatory shutdown and shunting in septic shock patients. In severe heart failure and cardiogenic shock, microcirculatory alterations are also frequently encountered and vasodilation may reverse this condition. Although the components of this treatment protocol are not innovative (and will also be available in the standard therapy group), guiding of this treatment by serial measurements of blood lactate levels is.

Intensive care extensively impacts on health care resources. Lactate-directed therapy aims at prevention of multiple organ failure (MOF) and subsequent death. Patients with MOF account for a disproportionately high part of the ICU budget. Moreover, in general costs per ICU day are higher for non-survivors than for survivors. Reduction in the use of ICU health care resources by lactate-directed therapy could thus result in an important economical benefit. In some hospitals, serial lactate measurements are routinely used on intensive care units. In our retrospective pilot study we found that in 2004 the Erasmus MC intensive care unit performed on average 12 lactate measurements per patient per admission. This resulted in a total of 28715 measurements with estimated external budget costs of € 336.000. If lactate-directed therapy appears equally or less effective than standard therapy, blood lactate measurement in the ICU may not be indicated and resources could thus be saved. Therefore, both a positive and negative outcome of this randomized controlled trial would be clinically and economically relevant.

The main research question of this study is, in patients with increased initial blood lactate levels on admission to the ICU:

1. will early lactate-directed therapy reduce mortality? (primary endpoint)
2. will early lactate-directed therapy reduce morbidity?
3. will early lactate-directed therapy reduce consumption of health care resources?

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the general ICU with an admission lactate level of ≥ 3,0 mmol/l
* Written informed consent

Exclusion Criteria:

* Liver failure
* Post liver surgery
* Age < 18 years
* Do not resuscitate status
* Contraindication to central venous or arterial catheterization
* Epileptic seizures (shortly before or during admission)
* Evident aerobic cause of hyperlactatemia
* Judgement of treating physician that study participation is undesirable for medical, medical-ethical or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2006-02; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality

SECONDARY OUTCOMES:
ICU mortality
Day-28 mortality
APACHE II,SOFA and hemodynamic variables
Use of health care resources
Pre-specified subgroup analyses within non-sepsis stratum:
Neuro critical care (traumatic brain injury, neurovascular conditions, neuro-oncological conditions)
Cardiac arrest
Remaining group (without neuro critical care and cardiac arrest)
Pre-specified subgroup analyses within sepsis stratum:
Sepsis and severe sepsis
Septic shock

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bakker, MD, PhD, Study Chair — Erasmus MC University Medical Center Rotterdam; Tim C Jansen, MD, Principal Investigator — Erasmus MC University Medical Center Rotterdam
Locations (5):
- Netherlands (5):
  - Reinier de Graaf Hospital, Delft
  - Erasmus MC University Medical Center, Rotterdam
  - Ikazia Hospital, Rotterdam
  - Medical Center Rijnmond Zuid, Rotterdam
  - St. Fransiscus Gasthuis, Rotterdam

REFERENCES:
- [Background] Retlich S, Duval V, Graefe-Mody U, Jaehde U, Staab A. Impact of target-mediated drug disposition on Linagliptin pharmacokinetics and DPP-4 inhibition in type 2 diabetic patients. J Clin Pharmacol. 2010 Aug;50(8):873-85. doi: 10.1177/0091270009356444. Epub 2010 Feb 16. PMID 20160157
- [Background] Williams DM, Jarrold C. Brief report: Predicting inner speech use amongst children with autism spectrum disorder (ASD): the roles of verbal ability and cognitive profile. J Autism Dev Disord. 2010 Jul;40(7):907-13. doi: 10.1007/s10803-010-0936-8. PMID 20112085
- [Background] Blow O, Magliore L, Claridge JA, Butler K, Young JS. The golden hour and the silver day: detection and correction of occult hypoperfusion within 24 hours improves outcome from major trauma. J Trauma. 1999 Nov;47(5):964-9. doi: 10.1097/00005373-199911000-00028. PMID 10568731
- [Background] Rossi AF, Khan DM, Hannan R, Bolivar J, Zaidenweber M, Burke R. Goal-directed medical therapy and point-of-care testing improve outcomes after congenital heart surgery. Intensive Care Med. 2005 Jan;31(1):98-104. doi: 10.1007/s00134-004-2504-1. Epub 2004 Dec 1. PMID 15650863
- [Background] Polonen P, Ruokonen E, Hippelainen M, Poyhonen M, Takala J. A prospective, randomized study of goal-oriented hemodynamic therapy in cardiac surgical patients. Anesth Analg. 2000 May;90(5):1052-9. doi: 10.1097/00000539-200005000-00010. PMID 10781452
- [Background] Levy B, Gibot S, Franck P, Cravoisy A, Bollaert PE. Relation between muscle Na+K+ ATPase activity and raised lactate concentrations in septic shock: a prospective study. Lancet. 2005 Mar 5-11;365(9462):871-5. doi: 10.1016/S0140-6736(05)71045-X. PMID 15752531
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Gozzoli V, Treggiari MM, Kleger GR, Roux-Lombard P, Fathi M, Pichard C, Romand JA. Randomized trial of the effect of antipyresis by metamizol, propacetamol or external cooling on metabolism, hemodynamics and inflammatory response. Intensive Care Med. 2004 Mar;30(3):401-7. doi: 10.1007/s00134-003-2087-2. Epub 2004 Jan 13. PMID 14722642
- [Background] Manthous CA, Hall JB, Olson D, Singh M, Chatila W, Pohlman A, Kushner R, Schmidt GA, Wood LD. Effect of cooling on oxygen consumption in febrile critically ill patients. Am J Respir Crit Care Med. 1995 Jan;151(1):10-4. doi: 10.1164/ajrccm.151.1.7812538.
- [Background] Bruder N, Lassegue D, Pelissier D, Graziani N, Francois G. Energy expenditure and withdrawal of sedation in severe head-injured patients. Crit Care Med. 1994 Jul;22(7):1114-9. doi: 10.1097/00003246-199407000-00011. PMID 8026200
- [Background] Raat NJ, Verhoeven AJ, Mik EG, Gouwerok CW, Verhaar R, Goedhart PT, de Korte D, Ince C. The effect of storage time of human red cells on intestinal microcirculatory oxygenation in a rat isovolemic exchange model. Crit Care Med. 2005 Jan;33(1):39-45; discussion 238-9. doi: 10.1097/01.ccm.0000150655.75519.02. PMID 15644646
- [Background] Spronk PE, Ince C, Gardien MJ, Mathura KR, Oudemans-van Straaten HM, Zandstra DF. Nitroglycerin in septic shock after intravascular volume resuscitation. Lancet. 2002 Nov 2;360(9343):1395-6. doi: 10.1016/s0140-6736(02)11393-6. PMID 12423989
- [Background] De Backer D, Creteur J, Dubois MJ, Sakr Y, Vincent JL. Microvascular alterations in patients with acute severe heart failure and cardiogenic shock. Am Heart J. 2004 Jan;147(1):91-9. doi: 10.1016/j.ahj.2003.07.006. PMID 14691425
- [Background] Moerer O, Schmid A, Hofmann M, Herklotz A, Reinhart K, Werdan K, Schneider H, Burchardi H. Direct costs of severe sepsis in three German intensive care units based on retrospective electronic patient record analysis of resource use. Intensive Care Med. 2002 Oct;28(10):1440-6. doi: 10.1007/s00134-002-1429-9. Epub 2002 Aug 17. PMID 12373469
- [Derived] Jansen TC, van Bommel J, Schoonderbeek FJ, Sleeswijk Visser SJ, van der Klooster JM, Lima AP, Willemsen SP, Bakker J; LACTATE study group. Early lactate-guided therapy in intensive care unit patients: a multicenter, open-label, randomized controlled trial. Am J Respir Crit Care Med. 2010 Sep 15;182(6):752-61. doi: 10.1164/rccm.200912-1918OC. Epub 2010 May 12. PMID 20463176